CLINICAL TRIAL: NCT05750329
Title: Clinical Study of Adjuvant Liver Transplantation Combined With Two-stage Hepatectomy for the Treatment of Patients With Unresectable Primary Hepatocellular Carcinoma, Colorectal Cancer With Liver Metastases, or End-stage Liver Disease: a Multicenter, Prospective, Single-arm Study
Brief Title: Liver Transplantation With Two-stage Liver Resection in Unresectable Liver Cancer , Metastases or Emd-stage Liver Disease (LTLR-LC)
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: RenJi Hospital (Other)
Collaborators: The Affiliated Hospital of Qingdao University (Other); The First Affiliated Hospital of Zhengzhou University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Renji-LT-2022-0001
Record Dates: First submitted 2023-01-04; First posted 2023-03-01 (Actual); Last update posted 2023-08-07 (Actual); Status verified 2023-08

CONDITIONS: Liver Transplant Disorder; Hepatic Cancer; End-stage Liver Disease
Keywords: liver transplantation; Hepatectomy
MeSH Terms: conditions — Liver Neoplasms; End Stage Liver Disease

STUDY DESIGN:
Intervention Model Description: All enrolled patients received assisted liver transplantation combined with two-stage hepatectomy Stage 1 Surgery: Left Hepatectomy, Left Lateral Graft Implantation, Portal Shunt to Graft Intermediate stage: continuous monitoring of liver function indexes and liver transplant donor volume after the first stage of surgery. Until the graft size reaches 0.8% of body weight (GBWR), or 35%-45% of the standard liver volume.
  Stage 2 Surgery: Residual Right Hepatectomy
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Surgical group (Experimental): All patients underwent left hepatectomy combined with orthotopic S2-3 liver segment transplantation, and then underwent autologous right hepatectomy after the graft had grown sufficiently large.
  Interventions: Procedure: assisted liver transplantation combined with two-stage hepatectomy

INTERVENTIONS:
Procedure: assisted liver transplantation combined with two-stage hepatectomy — Stage 1 Surgery: Left Hepatectomy, Left Lateral Graft Implantation, Portal Shunt to Graft Intermediate stage: continuous monitoring of liver function indexes and liver transplant donor volume after the first stage of surgery. Until the graft size reaches 0.8% of body weight (GBWR), or 35%-45% of the standard liver volume.
  Stage 2 Surgery: Residual Right Hepatectomy

SUMMARY:
Colon cancer and primary liver cancer are common malignant tumors with low survival rate worldwide, and unresectable primary liver cancer and colon cancer liver metastases have worse prognosis. End-stage liver disease is equated with advanced liver disease, liver failure and decompensated cirrhosis because they are generally irreversible. Liver transplantation is a treatment option for the above-mentioned patients and is expected to improve the prognosis of the patients, but the biggest problem faced by such patients is the shortage of donor livers. Recently, a new surgical modality, resection and partial liver segment 2-3 transplantation with delayed total hepatectomy (RAPID), can greatly alleviate these problems.Based on clinical surgical experience, our center proposes and designs a clinical study of adjuvant liver transplantation combined with two-stage hepatectomy in the treatment of patients with unresectable primary liver cancer, colorectal cancer liver metastases, or end-stage liver disease. By improvement of RAPID operation, the safety and efficacy of this treatment method in patients with those disease were evaluated.

ELIGIBILITY:
Inclusion Criteria:

1. aged 18-75 years;
2. patients with unresectable primary hepatocellular carcinoma or colorectal cancer with liver metastases who also meet the following criteria: tumor shrinkage (still unresectable) or no significant progression after a first-line chemotherapy regimen of 6-8 weeks; no other abdominal metastases or 1-3 resectable pulmonary metastases;
3. patients with end-stage liver disease;
4. preoperative Child classification of A or B, able to tolerate the subsequent surgical program
5. Signed informed consent Note: One of the second or third criteria needs to be fulfilled and all the rest of the selection criteria need to be fulfilled

Exclusion Criteria:

1. Extrahepatic tumor burden (except for resectable lung metastases) and/or macrovascular tumor infiltration
2. Tumor progression during chemotherapy or important comorbidities that affect surgery
3. Uncorrectable cardiopulmonary disease with high surgical risk
4. Anatomical abnormalities that preclude liver transplantation
5. Persistent non-compliance with medical care
6. Combined with other diseases such as AIDS that affect surgery or tumor progression

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-08 (Estimated); Primary Completion 2026-08 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Three-year overall survival rate after surgery | 3 years after the second liver resection
  After the second liver resection, patients were followed up through outpatient clinics and telephone (interval: once a month for a total of three years). The end point of follow-up was the death of the patient or survival after three years of follow-up. After reaching the end point of follow-up, the overall survival rate was analyzed by drawing survival curves.

SECONDARY OUTCOMES:
Postoperative tumor-free survival period | 3 years after the second liver resection
  After the second liver resection, regular follow-up of patients' serological and imaging indicators: Serological indicators include tumor markers, such as AFP, AFP heterogeneity, CEA, CA19-9, etc., imaging Medical indicators include abdominal ultrasound, enhanced CT, enhanced magnetic resonance or PET-CT examination. Serological examination and B-ultrasound examination should be performed once a month for the first year after surgery, and once every three months for the next two years. Enhanced CT or enhanced MRI should be performed at the 1st, 3rd, and 6th months after operation, and then once every six months (if the serology or B-ultrasound examination indicates abnormalities, an additional examination will be performed). Two or more imaging examinations diagnosed as malignant tumors were considered as tumor recurrence. Tumor recurrence or no recurrence after three years of follow-up was used as the end point of the study.